CLINICAL TRIAL: NCT05055284
Title: Efficacy of Patellar Taping and Electromyographic Biofeedback Training at Various Knee Angles on Quadriceps Strength and Functional Performance in Young Adult Male Athletes With Patellofemoral Pain Syndrome
Brief Title: Efficacy of Patellar Taping and Electromyographic Biofeedback Training at Various Knee Angles on Quadriceps Strength and Functional Performance in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU; IFP-2020-26 (Other Grant/Funding Number: Ministry of Education, Saudi Arabia)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Patellofemoral Disorder; Anterior Knee Pain Syndrome
Keywords: Pain; Strength; Function; PFPS; Athletes; SLTHT
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Experimental: Participants in this group will receive electromyography biofeedback (EMG-BF) guided strength training along with patellar taping at 30, 60, and 90-degree angles.
  No Intervention: Control: Participants in this group will receive Sham EMG-BF guided strength training without patellar taping at 30, 60, and 90-degree angles.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental: Participants in this group will receive electromyography biofeedback (EMG-BF) guided strength training along with patellar taping
  Interventions: Other: Electromyographic-biofeedback guided (EMG-BF) isometric quadriceps strengthening with patellar taping five days a week for six weeks.
- Control group (Sham Comparator): No Intervention: Control: Participants in this group will receive Sham EMG-BF guided strength training without patellar taping
  Interventions: Other: Electromyographic-biofeedback guided (EMG-BF) isometric quadriceps strengthening with patellar taping five days a week for six weeks.

INTERVENTIONS:
Other: Electromyographic-biofeedback guided (EMG-BF) isometric quadriceps strengthening with patellar taping five days a week for six weeks. — Patellar Taping, electromyography biofeedback (EMG-BF), Strength Training
  Other Names: Control group will receive Sham EMG-BF guided isometric quadriceps strengthening without patellar taping five days a week for six weeks.

SUMMARY:
This study compared the effects of patellar taping and electromyographic-biofeedback (EMG-BF) guided isometric quadriceps strengthening at different knee angles in patello-femoral pain syndrome (PFPS).

DETAILED DESCRIPTION:
A total of 60 adult male athletes aged 18 to 45 years were recruited. Subjects will be included with the history of knee pain during activities such as descending and ascending stairs, squatting, and running, had positive J sign (lateral tilt of patella), and a sign of patellar malalignment on the radiograph. Individuals with a history of fracture around the knee, patella dislocation, knee deformity (e.g., genu varum), flexion contracture, ligaments/meniscal injuries, and osteoarthritis of the knee will be excluded from the study. The protocol was submitted to and approved by the ethical sub-committee of the College of applied medical science, Majmaah, Saudi Arabia (Ethics number: MUREC-Nov./COM-2O20/11-2). Participants were requested to sign a written informed consent form approved by the institution ethics committee.

Participants were randomly assigned to Group A (experimental group): electromyography biofeedback (EMG-BF) guided maximum voluntary isometric contraction exercise with patellar taping; Group B (control group): sham EMG-BF guided maximum voluntary isometric contraction without patellar taping. The outcome measure for this study will be the mean changes in maximum voluntary isometric contraction (MVIC) of the quadriceps muscle at different angles, pain intensity, single-leg triple hop test (SLTH), and functional status up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain during activities such as descending and ascending stairs, squatting, and running,
* Positive J sign (lateral tilt of patella),
* Sign of patellar malalignment on the radiograph

Exclusion Criteria:

* Fracture around the knee,
* Patella dislocation,
* Knee deformity (e.g., genu varum),
* Knee flexion contracture,
* Ligaments/meniscal injuries, and
* Osteoarthritis of the knee.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Mean changes in pain intensity | 6 weeks
  The 10-cm visual analogue scale (VAS) will be used for the assessment of pain intensity. Each participant will be instructed to report their current intensity of pain on a 10-cm scale between two anchors 0 (indicates no pain) and 10 (indicates maximum pain).
Mean changes in knee function | 6 weeks
  Knee function will be assessed using the validated Anterior Knee Pain scale. It comprised of 13 questions designed to evaluate difficulties related to PFPS such as presence of a limp, walking ability, need for support, squatting, stair climbing, jumping, running, pain, abnormal painful kneecap movement, prolonged sitting with knees flexed, atrophy of the thigh, swelling, and flexion deficiency. Total scores range between 0 and 100. A higher score suggests lower symptoms and better functional capacity.
Mean changes in quadriceps muscle strength | 6 weeks
  Maximum voluntary isometric strength of quadriceps femoris muscle will be measured using an isokinetic dynamometer. Participants will be made in a sitting position and secured using the stabilization straps with the knee joint in 30,60,90 degrees of flexion, as this position has resulted in the most significant torque output. They will be verbally encouraged to carry out three maximal voluntary isometric contractions of quadriceps with 5-sec rest. The best of the three maximum peak torque will be used for the analysis.
Mean changes in balance performance | 6 weeks
  The SLTH test measured the distance participants travelled from the starting point to where the back of their heel touched the ground. They conducted three trials with a 3-minute rest period in between. The maximum distance covered score of the three, i.e., the best, was used as the baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan, PhD, Principal Investigator — Majmaah University
Locations (1):
- Physiotherapy & Rehabilitation center, Al Majma'ah, Riyadh Region, Saudi Arabia

REFERENCES:
- [Derived] Hasan S, Alonazi A, Anwer S, Jamal A, Parvez S, Alfaiz FAS, Li H. Efficacy of Patellar Taping and Electromyographic Biofeedback Training at Various Knee Angles on Quadriceps Strength and Functional Performance in Young Adult Male Athletes with Patellofemoral Pain Syndrome: A Randomized Controlled Trial. Pain Res Manag. 2022 Aug 1;2022:8717932. doi: 10.1155/2022/8717932. eCollection 2022. PMID 35958675